CLINICAL TRIAL: NCT00775697
Title: Montelukast Effects on Pulmonary Function in Children With Wheezing Aged Less Than 2 Years
Brief Title: Montelukast in Children With Wheezing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: Principal Investigator, Boner Attilio, Prof, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AABB1948
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Wheezing
Keywords: wheezing; children; montelukast; bronchodilators; lung function; Rint
MeSH Terms: conditions — Respiratory Sounds | interventions — montelukast; Leukotriene Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Montelukast (Experimental): the single arm will receive montelukast
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — the arm will be treated with Montelukast 4 mg die for 4 weeks
  Other Names: antileukotrienes
Drug: Montelukast — montelukast 4 mg day for 4 weeks
  Other Names: antileukotrienes

SUMMARY:
In this study children with recurrent wheezing (>/= 2 episodes in the last 6 months)and aged less than 2 years will be enrolled as outpatients. They will undergo lung function evaluation by Rint and by assessment of the flow curves at baseline and after 4 weeks of treatment with Montelukast 4 mg/day. Symptom dairies will be filled by parents during the study period.

DETAILED DESCRIPTION:
Patients aged less than 2 years with recurrent wheezing. At visit 1 patients with symptoms will be enrolled and the study explained. They will return home with bronchodilator therapy.

Within 1 week they will return for visit 2 to start a run-in period with bronchodilators prn and they will fill dairies with symptoms and drug use. Skin prick test will be evaluated at that time.

At visit 3 after 1 week of the run-in period they will start therapy with Montelukast 4 mg for 4 weeks, using bronchodilators prn and filling diaries.

The final visit will be after four weeks with re-evaluation of the lung function

ELIGIBILITY:
Inclusion Criteria:

* Age between 6-24 months
* Patients with recurrent wheezing (at least 2 episodes in the last 6 months)
* Patients with symptoms at enrollment

Exclusion Criteria:

* Chronic respiratory diseases (cystic fibrosis, chronic lung disease) symptoms at visit 1 that require hospital admission

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Lung function test (flow and resistance) | 4 weeks

SECONDARY OUTCOMES:
Bronchodilator use Dairy symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Attilio L Boner, MD, Principal Investigator — Universita di Verona
Locations (1):
- Clinica Pediatrica Universita' di Verona Policlinico GB Rossi, Verona, Italy